CLINICAL TRIAL: NCT02013609
Title: Protocol 331-13-003: An Exploratory, Multicenter, Open-label, Flexible-dose Trial of Brexpiprazole (OPC 34712) as an Adjunctive Treatment in Active Adults, 18 to 35 Years Old, With Major Depressive Disorder Who Are in a School or Work Environment.
Brief Title: Brexpiprazole (OPC-34712) as an Adjunctive Treatment in Active Adults, 18 to 35 Years Old, With Major Depressive Disorder Who Are in a School or Work Environment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-13-003
Record Dates: First submitted 2013-12-06; First posted 2013-12-17 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-02

CONDITIONS: MDD
Keywords: schizophrenia; Major depressive disorder; Anxiety Symptoms; School, Work environment; Mental Disorders; Psychotic Disorders; antipsychotic
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Anxiety Disorders; Mental Disorders; Psychotic Disorders | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brexpiprazole (Experimental): Up to 3mg/day, once daily dose, tablets, orally
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Treatment 12 weeks) - Up to 3 mg/day, once daily dose, tablets, orally

SUMMARY:
To investigate the efficacy and safety of flexibly dosed adjunctive brexpiprazole treatment in active adults with MDD, 18 to 35 years old, who are experiencing an inadequate selective serotonin reuptake inhibitor (SSRI)/serotonin norepinephrine reuptake inhibitor (SNRI) response in a school or work environment.

ELIGIBILITY:
Main Inclusion Criteria:

Have a diagnosis of a single or recurrent, nonpsychotic episode of MDD as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) and confirmed by both the Mini International Neuropsychiatric Interview (M.I.N.I.) and an adequate clinical psychiatric evaluation.

Have a treatment history of an inadequate ADT response to at least 1 ADT (but not > 3) for the current episode.

Have received a single, trial-approved, SSRI or SNRI at an adequate dose for ≥ 6 weeks prior to screening.

Are 18 to 35 years old at the time of consent (inclusive, and outpatients only).

Are (and will be) working 20 hours or more per week or a student taking 6 credit hours or more during the trial period, however minor deviations from the "part-time" concept may be acceptable on a case-by-case basis based on approval of the medical monitor.

Have a Hamilton Depression Rating Scale (HAM-D)- 17-item Total Score ≥ 18 at screening and baseline.

Have a Sheehan Disability Scale (SDS) 3-item mean score ≥ 5 at baseline.

Main Exclusion Criteria:

Subjects with any of the following current Axis I DSM-IV-TR diagnoses: delirium, dementia, amnestic, or other cognitive disorders; schizophrenia, schizoaffective disorder, or other psychotic disorders; bipolar I disorder, bipolar II disorder, or bipolar disorder not otherwise specified (NOS); eating disorders (including anorexia nervosa or bulimia); obsessive compulsive disorder; panic disorder; post-traumatic stress disorder; and attention deficit hyperactivity disorder.

Subjects with any of the following current Axis II DSM-IV-TR diagnoses: borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorders, or mental retardation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junichi Hashimoto, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd Japan (OPCJ)
Locations (24):
- United States (24):
  - Cerritos, California
  - Costa Mesa, California
  - Garden Grove, California
  - Glendale, California
  - Orange, California
  - Riverside, California
  - San Diego, California
  - Norwich, Connecticut
  - Fort Myers, Florida
  - Hialeah, Florida
  - Melbourne, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Prairie Village, Kansas
  - Weymouth, Massachusetts
  - Las Vegas, Nevada
  - Brooklyn, New York
  - Jamaica, New York
  - Staten Island, New York
  - Portland, Oregon
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Seattle, Washington

REFERENCES:
- [Derived] Weiss C, Meehan SR, Brown TM, Gupta C, Morup MF, Thase ME, McIntyre RS, Ismail Z. Effects of adjunctive brexpiprazole on calmness and life engagement in major depressive disorder: post hoc analysis of patient-reported outcomes from clinical trial exit interviews. J Patient Rep Outcomes. 2021 Dec 11;5(1):128. doi: 10.1186/s41687-021-00380-4. PMID 34894307

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 48 participants at 24 sites in the United States; 15 of the 24 trial sites enrolled participants.
Pre-assignment Details: The trial consisted of a 2 to 21-day screening phase, a 12-week (84-day) treatment phase, and a 30-day (+ 2) follow-up phase.
Groups:
- Brexpiprazole: Participants were administered oral brexpiprazole tablet of 0.5 milligram per day (mg/day) for the first week with titration up to 3 mg/day once daily (QD) in addition to their constant-dose antidepressant therapy (ADT) for 12 weeks.
Period: Overall Study
Arm/Group | Brexpiprazole
Started | 47 (One participant out of 48 participants enrolled had discontinued before receiving study medication.)
Completed | 29
Not Completed | 18
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 3
Not completed — Met Withdrawal Criteria | 3

BASELINE CHARACTERISTICS:
Groups:
- Brexpiprazole: Participants were administered oral brexpiprazole tablet of 0.5 mg/day for the first week with titration up to 3 mg/day QD in addition to their constant-dose ADT for 12 weeks.
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 12 in the Montgomery Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS was utilized as the primary efficacy assessment of the participant's level of depression and was administered utilizing the Structured Interview Guide for the MADRS (SIGMA). Detailed instructions for administration of this structured interview was provided in the SIGMA. The MADRS consists of 10 items, all rated on a 0 to 6 scale with 0 being the "best" rating and 6 being the "worst" rating. The MADRS Total Score is the sum of ratings for all 10 items. The possible Total scores are from 0 to 60.
Time Frame: Baseline and Week 12
Population: All participants who took at least one dose of brexpiprazole and who had a valid Baseline assessment and at least one valid Post-Baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
Units on a scale | -18.1 (1.4)
Statistical Analysis 1: Comparison: Brexpiprazole; The null hypothesis of zero in mean change from Baseline in MADRS total score at Week 12 was tested at significance level of 0.05. Since this is an exploratory trial, no methods to control type I error rate were performed; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed model repeated measure (MMRM) with model terms: Baseline, visit, and Baseline by visit interaction

2. Secondary Outcome: Mean Change From Baseline to Week 12 in Clinical Global Impression-Severity (CGI-S) Total Score
Description: The severity of illness for each participant was rated using the CGI-S. To perform this assessment, the study physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
Units on a scale | -2.0 (0.2)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM with model terms: Baseline, visit, and Baseline by visit interaction

3. Secondary Outcome: Mean Clinical Global Impression-Improvement (CGI-I) Score at Week 12
Description: The improvement of each participants condition was rated for each participant using the CGI-I. The study physician rated the participants total improvement whether or not it was due entirely to drug treatment. To perform this assessment, the study physician answered the following question: "Compared to his/her condition at baseline, how much has the participant changed?" Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. The response at a given week was compared with the participants condition at Baseline prior to the first dose of study medication.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 8, 10 and 12
Population: Participants who took at least 1 dose of brexpiprazole with a valid Baseline assessment and at least one valid Post-Baseline efficacy assessment; the last-observation-carried-forward (LOCF) dataset included data recorded at a scheduled visit or, data was carried forward from the previous scheduled visit, if no observation was recorded at that visit
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
Units on a scale
  Week 1 (N= 46) | 3.5 (0.8)
  Week 2 (N= 47) | 3.0 (0.8)
  Week 3 (N= 47) | 2.8 (1.0)
  Week 4 (N= 47) | 2.7 (1.0)
  Week 6 (N= 47) | 2.6 (1.3)
  Week 8 (N= 47) | 2.5 (1.2)
  Week 10 (N= 47) | 2.3 (1.2)
  Week 12 (N= 47) | 2.2 (1.3)

4. Secondary Outcome: Number of Participants With CGI-I Response
Description: The CGI-I response rate was defined as a CGI-I score of 1 (very much improved) or 2 (much improved).
Time Frame: Weeks 1, 2, 3, 4, 6, 8 ,10 and 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
participants
  Week 1 (N= 46) | 4
  Week 2 (N= 47) | 12
  Week 3 (N= 47) | 17
  Week 4 (N= 47) | 24
  Week 6 (N= 47) | 27
  Week 8 (N= 47) | 29
  Week 10 (N= 47) | 28
  Week 12 (N= 47) | 30

5. Secondary Outcome: Percentage of Participants With MADRS Response
Description: MADRS response rate was defined as ≥ 50% reduction in respective total scores from Baseline to Week 12.
Time Frame: Baseline and Week 12
Population: Participants who took at least 1 dose of brexpiprazole with a valid Baseline assessment and at least one valid Post-Baseline efficacy assessment. The LOCF data set included data recorded at a scheduled treatment phase visit or, data was carried forward from the previous scheduled treatment phase visit, if no observation was recorded at that visit.
Measure: Number; unit: percentage of particpants
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
percentage of particpants | 53.2

6. Secondary Outcome: Percentage of Participants With MADRS Remission
Description: MADRS remission rate, where remission is defined as MADRS Total Score ≤ 10 and 50% reduction in MADRS Total Score from Baseline to Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
percentage of participants | 42.6

7. Secondary Outcome: Mean Change From Baseline to Week 12 in Hamilton Depression Rating Scale (HAM-D17) Total Score
Description: The HAM-D17 was utilized as an assessment of a participants level of depression and was administered utilizing the Structured Interview Guide for the Hamilton Depression Rating Scale (SIGH-D). Detailed instructions for administration of this structured interview were provided in the SIGH-D. HAM-D17 is a 17-item questionnaire with a total score of 0 to 52 with higher scores indicating more depressive symptoms.
Time Frame: Baseline and Week 12
Population: All participants who took at least one dose of brexpiprazole and who had a valid Baseline assessment and at least one valid Post-Baseline efficacy assessment. Mixed model repeated measures was performed on the OC dataset.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
Units on a scale | -14.9 (1.1)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM with model terms: Baseline, visit, and Baseline by visit interaction

8. Secondary Outcome: Mean Change From Baseline to Week 12 in Sheehan Disability Scale (SDS) 3-item Total/Summed Score
Description: The SDS was a self-rated instrument used to measure the effect of the participant's symptoms on work/school, social life, and family/home responsibilities. The SDS was a visual analogue scale that used spatio-visual, numeric, and verbal descriptive anchors simultaneously to assess disability across the 3 domains. The number most representative of how much each area was disrupted by symptoms was marked along the line from 0 = not at all to 10 = extremely. Scores of 5 and above were associated with significant functional impairment. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired).
Time Frame: Baseline and Week 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
Units on a scale | -3.74 (0.54)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM with model terms: Baseline, visit, and Baseline by visit interaction

9. Secondary Outcome: Mean Change From Baseline to Week 12 in Sheehan Disability Scale (SDS) Single Item Sub-scores
Description: The SDS was a self-rated instrument used to measure the effect of the participant's symptoms on work/school, social life, and family/home responsibilities. The SDS was a visual analogue scale that used spatio-visual, numeric, and verbal descriptive anchors simultaneously to assess disability across the 3 domains. The number most representative of how much each area was disrupted by symptoms was marked along the line from 0 = not at all to 10 = extremely. Scores of 5 and above were associated with significant functional impairment.
Time Frame: Baseline and Week 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
Units on a scale
  Work/ school | -3.5 (0.5)
  Social life | -3.9 (0.6)
  Family life/ home responsibilities | -3.7 (5.0)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12 of single item sub-scores of tasks: work/ school, social life and family life/ home responsibilities; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — The p-value is the same for each of single item sub-scores of tasks: work/ school, social life and family life/ home responsibilities; MMRM with model terms: Baseline, visit, and Baseline by visit interaction

10. Secondary Outcome: Mean Change From Baseline to Week 12 in Social Adaptation Self-evaluation Scale (SASS) Total Score
Description: The SASS was a self-rated instrument to assess the social motivation and behavior in participants with depression. It contained 21 items covering the different aspects of social interactions, global social attitude, and self-perception. The SASS total score will be un-evaluable if less than 16 of the 20 items (for item number 1 and item number 2, participant is to answer either one of these) are recorded. If 16 to 19 of the 20 items are recorded, the SASS total score will be the mean of the recorded items multiplied by 20 and then rounded to the first decimal place.Each item is scored from 0 to 3, corresponding to minimal and maximal social adjustment, with a total score range of 0 to 60 (higher scores, indicating worse outcome).
Time Frame: Baseline and Week 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
Units on a scale | 9.7 (1.6)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM with model terms: Baseline, visit, and Baseline by visit interaction

11. Secondary Outcome: Mean Change From Baseline to Week 12 in Massachusetts General Hospital-Cognitive and Physical Functioning Questionnaire (MGH-CPFQ) Total Score
Description: The MGH-CPFQ was a participant-rated scale designed to assess cognitive and executive dysfunction including symptoms of fatigue in mood and anxiety disorders. The MGH-CPFQ consisted of 7 items, each rated on a scale from 1 (greater than normal functioning) to 6 (poorer than normal functioning). The total score of the 7 items ranged from 7 to 42.
Time Frame: Baseline and Week 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
Units on a scale | -8.1 (1.3)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM with model terms: Baseline, visit, and Baseline by visit interaction

12. Secondary Outcome: Mean Change From Baseline to Week 12 in Kellner Symptom Questionnaire (KSQ) Total Score
Description: KSQ is a subject-rated scale designed to assess distress using symptoms of depression, anxiety, anger-hostility and somatization. The questionnaire contains 92 items of which 68 items indicate symptoms and 24 items are antonyms of some of the symptoms that indicate well-being. The maximum score for each symptom subscale is 17, the well-being subscales 6 and for the total scale scores 23.The total subscale scores will be unevaluable if less than 19 of the 23 items are recorded. If 19 to 22 of the 23 items are recorded, the total subscale score is the mean of the recorded items multiplied by 23 and then rounded to the first decimal place. The total score will be unevaluable if less than 76 of the 92 items are recorded. If 76 to 91 of the 92 items and no less than 19 of the 23 items of each subscale are recorded, the total score will be the mean of the recorded items multiplied by 92 and then rounded to the first decimal place. A higher score indicates more distress than a lower score.
Time Frame: Baseline and Week 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
Units on a scale | -30.5 (3.6)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM with model terms: Baseline, visit, and Baseline by visit interaction

13. Secondary Outcome: Mean Change From Baseline to Week 12 in Go/No-Go Task (P-inhibition Failure)
Description: Executive function and working memory were assessed for the Go/No-go Task using computer-based and paper-pencil neuropsychological instruments. These instruments focused on measuring impulse inhibition. Proportions of inhibitory failures (p-inhibitory failures) is measured as the proportion of no-go targets in the go-cue condition in which a participant failed to inhibit a response.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: failures
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 45
failures
  P-inhibition failures (Go cues) | 0.052 (0.299)
  P-inhibition failures (No-Go cues) | 0.052 (0.295)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12 for p-inhibition failures (Go cues); Test type: Superiority or Other; p = 0.3439, t-test, 2 sided; p-value for change from Baseline using t-test
Statistical Analysis 2: Comparison: Brexpiprazole; Statistical analysis at Week 12 for p-inhibition failures (No-Go cues); Test type: Superiority or Other; p = 0.3385, t-test, 2 sided; p-value for change from Baseline using t-test

14. Secondary Outcome: Mean Change From Baseline to Week 12 in Go/No-Go Task (Mean Reaction Time)
Description: Executive function and working memory were assessed for the Go/No-go Task using computer-based and paper-pencil neuropsychological instruments. These instruments focused on measuring impulse inhibition.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 45
milliseconds
  Mean reaction time (Go cues) | -17.35 (73.34)
  Mean reaction time (No-Go cues) | -12.99 (70.67)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12 for mean reaction time (Go cues); Test type: Superiority or Other; p = 0.2052, t-test, 2 sided; p-value for change from Baseline using t-test
Statistical Analysis 2: Comparison: Brexpiprazole; Statistical analysis at Week 12 for mean reaction time (No-Go cues); Test type: Superiority or Other; p = 0.3224, t-test, 2 sided; p-value for change from Baseline using t-test

15. Secondary Outcome: Mean Change From Baseline in Delay Discounting Task - Monetary Choice Questionnaire (MCQ) k Value
Description: Delay discounting was a participant-completed task is an index of impulsive behavior. It measured the extent to which the value of a reward decreased as the delay to obtaining that reward increased. The propensity of participants to delay reward was assessed with an MCQ. Discounting rate is estimated using, k= (A/V)1/D, where k is the discounting rate parameter, V is the immediate reward, A is the higher delayed reward and D is the amount of days to the delayed reward. The MCQ consists of 27 choices between immediate and delayed rewards. The participant chooses repeatedly between 2 hypothetical sums of money: a smaller amount now or a larger amount in the future (for example, "would you prefer $27 today or $50 in 21 days?") The answers provide an estimate of the participant's discounting rate; higher discounting rates indicate greater impulsivity. A total score is not computed for all 27 questions.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
unitless | 0.009531 (0.055516)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.3169, t-test, 2 sided; p-value for change from Baseline using t-test

16. Secondary Outcome: Mean Change From Baseline to Week 12 in the Number of Impulsive Choices in the Delayed Reward Task (DRT)
Description: Delay discounting was a participant-completed task considered as an index of impulsive behavior. It measured the extent to which the value of a reward decreased as the delay to obtaining that reward increased. During a training session, a single button with letter A or B appeared on the screen. The participant had to wait until the letter began to flash, and press the button only once. An amount of money was added to a counter and another single button appeared. During the test session, both buttons with letters A and B appeared on the screen. The participant had to choose one of the letters that remained; the other disappeared. The participant had to wait until the letter began to flash and then press the button again. An amount of money was added to the counter, and both letters appeared again. The data are computerized and reflect delay discounting and impulsivity (higher discounting shows greater impulsivity). A total score was not calculated for this task.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Number of Impulsive Choices
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 37
Number of Impulsive Choices | 3.6 (15.2)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.3352, t-test, 2 sided

17. Secondary Outcome: Mean Change From Baseline to Week 12 in Delay and Probability Discounting Task (DPDT)
Description: The experiential discounting task (EDT) was a subject-completed computerized task designed to measure delay discounting, an index of impulsive behavior. It measured the extent to which the value of a reward decreased as the delay to obtaining that reward increased. The participant chose between different amounts of money available at different delays or with different chances (probability to get the money). At the end of the session, one of the choices was selected at random, and the participant received whatever they chose in response of that question (immediate, delayed, or probabilistic amount). Formula for h-value:value = A / (1 + hO) p is probability of reward and O is odds against.The value of h indicates how the value of a reward and the probability of its occurrence decreases.The data are computerized and reflect delay discounting and impulsivity (higher discounting and higher probability discounting shows greater impulsivity). A total score is not computed for this task.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 41
unitless
  Delay Discounting Task k value | 21.315241 (116.798133)
  Delay Discounting Task h value | 10.350419 (60.212518)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12 for delay discounting task k value; Test type: Superiority or Other; p = 0.3517, t-test, 2 sided
Statistical Analysis 2: Comparison: Brexpiprazole; Statistical analysis at Week 12 for delay discounting task h value; Test type: Superiority or Other; p = 0.3799, t-test, 2 sided

18. Secondary Outcome: Mean Change From Baseline in Food Delay Discounting Task (DDT)
Description: Delay discounting was a participant-completed task considered as an index of impulsive behavior. The participant chooses between a reward they could have today and another that they could get after a specified amount of time. The participant would not receive the rewards, but was asked to make decisions as though he or she were really going to receive them. AUC is defined as area under the concentration-time curve; AUC for food is presented below. The data are computerized and reflect delay discounting and impulsivity (higher discounting shows greater impulsivity). To calculate the AUC, the "X-axis" is "days", "Y-axis" is "Food value", the actual area underneath the curve was calculated by summing the results for each delay and present value pair: x2 -x1[(y1 + y2)/2], where x1 and x2 are successive delays and y1 and y2 are the present values associated with those delays. The AUC can range from 1 (no discounting) to 0 (maximum discounting).
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 30
unitless | 0.3487 (1.4158)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12 (AUC for food); Test type: Superiority or Other; p = 0.2610, t-test, 2 sided
Statistical Analysis 2: Comparison: Brexpiprazole; Statistical analysis at Week 12 (AUC for money); Test type: Superiority or Other; p = 0.8138, t-test, 2 sided

19. Secondary Outcome: Mean Change From Baseline in Money Delay Discounting Task
Description: Delay discounting was a participant-completed task considered as an index of impulsive behavior. The participant chose between a reward they could have today and another that they could get after a specified amount of time. The participant would not receive the rewards, but was asked to make decisions as though he or she were really going to receive them. AUC is defined as area under the concentration-time curve; AUC for money is presented below. The data are computerized and reflect delay discounting and impulsivity (higher discounting shows greater impulsivity). To calculate the AUC, the "X-axis" is "days", "Y-axis" is "Money value", the actual area underneath the curve was calculated by summing the results for each delay and present value pair: x2 -x1[(y1 + y2)/2], where x1 and x2 are successive delays and y1 and y2 are the present values associated with those delays. The AUC can range from 1 (no discounting) to 0 (maximum discounting).
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 30
unitless | -0.0095 (0.1859)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12 (AUC for money); Test type: Superiority or Other; p = 0.8138, t-test, 2 sided

20. Secondary Outcome: Mean Change From Baseline to Week 12 in Barratt Impulsiveness Scale 11-Item (BIS-11) Total Score
Description: The BIS-11 was a participant-rated scale designed to assess impulsive personality traits. The BIS-11 consisted of 30 items scored on a 4-point scale ranging from 1 (rarely/never) to 4 (almost always/always). The scores provided information to assess 6 first-order factors (attention, motor, self-control, cognitive complexity, perseverance, and cognitive instability impulsiveness) and 3 second-order factors (motor impulsiveness, non-planning impulsiveness, and attentional impulsiveness). The total score ranged from 30 to 120, with higher scores indicating impulsive personality traits.
Time Frame: Baseline and Week 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
Units on a scale | -7.1 (1.5)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis at Week 12; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM with model terms: Baseline, visit, and Baseline by visit interaction

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of the informed consent until the last dose of brexpiprazole with a safety follow-up of 30 (+2) days.
Description: One participant out of 48 participants enrolled had discontinued before receiving study medication.
Arm/Group | Brexpiprazole
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 39/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=47)
Abdominal Discomfort (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 5
Weight increased (Investigations) | 8
Increased appetite (Metabolism and nutrition disorders) | 3
Akathisia (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 10
Sedation (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 8
Anxiety (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 5
Libido decreased (Psychiatric disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No